CLINICAL TRIAL: NCT05951621
Title: Effect of Qigong on Gestational Diabetes Mellitus：A Randomized Controlled Trial
Brief Title: The Patients With Gestational Diabetes Were Interfered With Qigong.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chen Chaoyang (Other)
Collaborators: Shanghai First Maternity and Infant Hospital (Other)
Responsible Party: Sponsor-Investigator, Chen Chaoyang, Shanghai Qigong Research Institute Trainee researcher, Shanghai University of Traditional Chinese Medicine
Organization: Shanghai University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZY(2021-2023)- 0105-14
Record Dates: First submitted 2023-07-11; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy
Keywords: Gestational Diabetes Mellitus in Pregnancy; Qigong; Non-drug therapy
MeSH Terms: interventions — Qigong; Exercise

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Qigong group (Experimental): On the basis of nutrition and exercise management and guidance, Qigong is exercised. Offline intensive learning once a week, 45-60 minutes each time, study for 12 weeks, and arrange online theory lecture once a week. In addition to concentrated learning, subjects in this group were required to practice themselves at home, at least once a day, each time for 30 minutes.
  Interventions: Other: Qigong
- Control group (Experimental): guidance of nutrition and exercise
  Interventions: Behavioral: guidance of nutrition and exercise

INTERVENTIONS:
Other: Qigong — An ancient Chinese system of postures, exercises, breathing techniques, and meditations designed to improve and enhance the body's QI.
  Arms: Qigong group
Behavioral: guidance of nutrition and exercise — Provide health promotion and guidance to participants on diet and physical exercise
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to learn about in women with gestational diabetes's health conditions.

The main question[s] it aims to answer are:

* Can Qigong control blood glucose in women with gestational diabetes?
* Can Qigong improve mood and sleep in women with gestational diabetes? Participants will required to follow the research team for 3 months of qigong practice。 If there is a comparison group: Researchers will compare Qigong groups to see if Qigong's effects.

ELIGIBILITY:
Inclusion Criteria:

* 20 years old≤ age ≤ 40 years old;
* Those with clear awareness, acceptable reading and language expression skills, and barrier-free communication;
* singleton pregnancy;
* gestational age between 24 and 28 weeks, with the upper limit of gestational age set at 28 weeks at the time of inclusion to allow for at least 8 weeks of intervention;
* Body mass index (BMI) is lower than 40;
* Agree to participate in this project and sign the informed consent form.

Exclusion Criteria:

* Those with previous GDM and diabetes;
* Artificial insemination;
* Those with serious obstetric complications and contraindications;
* Participants in other planned and supervised exercise programs or researchers during the study.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Fasting blood glucose | Average peripheral fasting blood glucose measured one week prior to participant enrollment. Fasting blood glucose measured in the first week after the end of 12 weeks of intervention.
  If the blood glucose level is between 4.0 and 5.4 mmol/L, the result is normal. If the fasting blood glucose level is between 5.5-6.9 mmol/L, the condition is called prediabetes. Diabetes refers to blood sugar greater than 8.5 mmol/L.
2-h postprandial plasma glucose | Average postprandial blood glucose measured in the week prior to study participant enrollment. Average postprandial 2-hour postprandial peripheral capillary blood glucose measured in the first week after the end of 12 weeks of intervention.
  less than 7.8mmol/L. When the blood glucose is 7.8~11.1 mmol/L 2 hours after meals, it can be diagnosed as impaired or impaired glucose tolerance.

SECONDARY OUTCOMES:
Pittsburgh sleep quality index,PSQI | Weeks 0 and 13
  PSQI was used to measure the sleep quality of participants in the last 1 month. It consists of 19 self-assessment items and 5 other assessment items, of which the 19th self-assessment item and 5 other evaluation items do not participate in scoring, and only 18 self-assessment items participating in scoring are introduced here. 18 items composed of 7 components, each component is scored on a scale of 0-3, the cumulative score of each component is the total score of PSQI, the total score range is 0-2l, the higher the score, the worse the sleep quality.
Self-Rating Depression Scale，SDS | Weeks 0 and 13
  SDS is rated according to the frequency of symptoms and is divided into 4 levels: no or very little time, a small amount of time, a considerable amount of time, and most or all the time. If it is a positive scoring question, it is rated as a rough score of L, 2, 3, and 4. For reverse grading questions, they are rated as 4, 3, 2, and 1. The assessment time is within the past week, add the scores of each question to a rough score, multiply the rough score by 1.25, and round up the whole number to get the standard score (T). The threshold value of depression assessment is T=53, and the higher the score, the more obvious the tendency to depression.
Self-Rating Anxiety Scale, SAS | Weeks 0 and 13
  SAS includes 20 items, and the score is based on a standard scoring pattern, with a score of 50 or less being normal, 50-59 being mild anxiety, 60-69 being moderate anxiety, and 70-79 being severe anxiety.

OTHER OUTCOMES:
Maternal and infant complications during childbirth | birth

CONTACTS AND LOCATIONS:
Overall Officials: Li Jie, Doctor, Principal Investigator — Shanghai University of Traditional Chinese Medicine

IPD SHARING:
Plan to Share IPD: No
This study is still in the exploratory stage and has a certain degree of confidentiality

REFERENCES:
- [Background] Jin Y, Chen Z, Li J, Zhang W, Feng S. Effects of the original Gymnastics for Pregnant Women program on glycaemic control and delivery outcomes in women with gestational diabetes mellitus: A randomized controlled trial. Int J Nurs Stud. 2022 Aug;132:104271. doi: 10.1016/j.ijnurstu.2022.104271. Epub 2022 Apr 28. PMID 35660387
- [Background] Sklempe Kokic I, Ivanisevic M, Biolo G, Simunic B, Kokic T, Pisot R. Combination of a structured aerobic and resistance exercise improves glycaemic control in pregnant women diagnosed with gestational diabetes mellitus. A randomised controlled trial. Women Birth. 2018 Aug;31(4):e232-e238. doi: 10.1016/j.wombi.2017.10.004. Epub 2017 Oct 18. PMID 29055674
- [Background] Yew TW, Chi C, Chan SY, van Dam RM, Whitton C, Lim CS, Foong PS, Fransisca W, Teoh CL, Chen J, Ho-Lim ST, Lim SL, Ong KW, Ong PH, Tai BC, Tai ES. A Randomized Controlled Trial to Evaluate the Effects of a Smartphone Application-Based Lifestyle Coaching Program on Gestational Weight Gain, Glycemic Control, and Maternal and Neonatal Outcomes in Women With Gestational Diabetes Mellitus: The SMART-GDM Study. Diabetes Care. 2021 Feb;44(2):456-463. doi: 10.2337/dc20-1216. Epub 2020 Nov 12. PMID 33184151
- [Background] Brown J, Ceysens G, Boulvain M. Exercise for pregnant women with gestational diabetes for improving maternal and fetal outcomes. Cochrane Database Syst Rev. 2017 Jun 22;6(6):CD012202. doi: 10.1002/14651858.CD012202.pub2. PMID 28639706